CLINICAL TRIAL: NCT05646173
Title: Comparison of the Efficacy of Auricular Vagus Nerve Stimulation and Electrotherapy Modalities in Chronic Low Back Pain
Brief Title: Efficacy of Auricular Vagus Nerve Stimulation and Electrotherapy Modalities in Patients With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: low back pain
Record Dates: First submitted 2022-10-18; First posted 2022-12-12 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2022-10

CONDITIONS: Low Back Pain
Keywords: vagus nerve stimülation
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: 60 patients, aged between 18 and 60, with persistent low back pain who voluntarily agreed to participate in the study will be included in the study. Patient Identification Form, Lumbal Region Joint Range of Motion and Mobility (Inclinometer, Modified Schober Test), muscle strength (CSMI-Cybex Humac-Norm isokinetic dynamometer and manual muscle strength measuring device) in the evaluation of patients with CKD and endurance tests, postural control and balance assessment (BBS, Biodex Medical Systems), Visual Analogue Scale (VAS), Beck Depression Inventory (BDI), Pittsburgh Sleep Quality Scale (PUKÖ), Oswestry Disability Index. Statistical analysis will be calculated using SPSS for Windows 22 program.
Masking Description: Double (Participant, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- grup 1 (Active Comparator): Grup 1: Participants will be treated with ultrasound (5 min), TENS with a hot pack for (20 minutes). Home exercises will be given. The home exercises will be given consist of isometric waist, hip flexor stretching, hamstring stretching, self-mobilization exercise, waist and abdominal concentric strength exercises.
  1.5w/cm² continuous ultrasound wiil applied with Chattanooga Intelect Mobile Ultrasound device.TENS: It will be applied to the lumbar region with a COMPEX brand stim device, together with a hot pack.The current intensity was opened by questioning according to the sensory threshold of the people.
  Home based exercise program:In the first week of the exercise program; isometric exercises, stretching and mobilization exercises were given. Second week; additional bridging exercise; In the third week, additional isotonic, active abdominal and back strengthening exercises were included in all exercises.
  The application will be done in 15 sessions, 5 days a week
  Interventions: Device: Electrophysical agents; Other: home exercise program
- grup 2 (Experimental): Grup 2: Participants will be given auricular vagus stimulation (25 min). Home exercises will be given. The home exercises will be given consist of isometric waist, hip flexor stretching, hamstring stretching, self-mobilization exercise, waist and abdominal concentric strength exercises.
  Vagus stimulation: A specially manufactured earphone that can be selected according to the size of the ear placed in the outer ear will be applied from the vagustim device (frequency 10 Hz, pulse duration less than 500 microseconds, in modulated TENS mode and biphasic asymmetric waveform) connected to it.
  Home based exercise program: In the first week of the exercise program; isometric exercises, stretching and mobilization exercises were given. Second week; additional bridging exercise; In the third week, additional isotonic, active abdominal and back strengthening exercises were included in all exercises.
  The application will be done in 15 sessions, 5 days a week.
  Interventions: Device: vagus stimülation device; Other: home exercise program

INTERVENTIONS:
Device: vagus stimülation device — Vagustim is a wearable medical technology device that focuses on non-invasive bilateral auricular vagus nerve stimulation (VNS). VNS is a clinically approved, safe and effective neuromodulation method.
  Arms: grup 2
Device: Electrophysical agents — Electrophysical agents (EPAs) are those modalities that administer thermal, mechanical, electrical or light energy to the patient to provide physiological effects and therapeutic benefits.
  Arms: grup 1
Other: home exercise program — The home exercise program will be explained to the patients by the physiotherapist and will also be given to the patient in the form of a brochure. Patients will be instructed to do the exercises regularly, three times a day for ten repetitions each day. The content of the exercises is updated weekly.

SUMMARY:
The aim of our study is to compare the effectiveness of auricular vagus nerve stimulation and conventional physical therapy in patients with Chronic Low Back Pain (CBA). 60 patients, aged between 18 and 60, with persistent low back pain for the last 3 months and who voluntarily agreed to participate in the study will be included in the study. Patients will be randomly divided into two groups as conventional therapy (Group I) and auricular vagus stimulation therapy (Group II). Patient Identification Form, Oswestry Disability Index, Lumbal Region Joint Range of Motion and Mobility (Inclinometer, Modified Schober Test, Hand Finger-Ground Distance Test), muscle strength (CSMI-Cybex Humac-Norm isokinetic dynamometer and Lafayette manual muscle strength measuring device) in the evaluation of patients with CKD and endurance tests, postural control and balance assessment (BBS, Biodex Medical Systems), Visual Analogue Scale (VAS), Beck Depression Inventory (BDI), Pittsburgh Sleep Quality Scale (PUKÖ). After the measurements on the 1st day, 15 sessions of application and the measurements will be repeated the day after the last session. A home exercise program will be created for the patients in both groups. Statistical analysis will be calculated using SPSS for Windows 22 program.

DETAILED DESCRIPTION:
Low back pain is one of the common problems that 80% of people experience at least once in their lifetime. Treatment of chronic low back pain includes surgical treatment, medical treatment and conservative treatment. The aim of conservative treatment is to raise the patient to the best possible level. Evidence levels for approaches commonly used in the clinic for the treatment of chronic low back pain were generally very low to moderate. It has been stated that the success of treatment is low in patients who are taken to conventional rehabilitation in the clinic, due to the lack of personal programs and the problems caused by the lack of human resources and space.

In recent studies, it has been shown that vagal nerve stimulation modulates peripheral and central nociceptive functions and reduces pain response. As a result, it was found that the pain threshold increased and the mechanical pain sensitivity decreased.

When we look at the literature; Although there are many studies on the treatment of chronic low back pain, there are no studies on the use of vagus nerve stimulation. Vagus nerve stimulation can be used as an adjunct therapy to correct autonomic nerve dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* be between the ages of 20-60
* volunteering to work
* Having low back pain for more than 3 months
* Diagnosis of chronic low back pain by the doctor
* Being able to read and write and be cooperative.
* Not having received treatment for the lumbar region in the last 3 months

Exclusion Criteria:

* Not having any lumbar surgery or vertebral fracture
* Being neurological, radiculopathy, inflammatory etc disease
* Having spinal deformities such as scoliosis or kyphosis
* Vestibular or respiratory disorder, Auditory or cognitive impairment
* Taking medication that will affect the balance (sedatives, etc.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2023-02-08 (Actual); Study Completion 2023-03-27 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODİ) | 3 week
  The Oswestry Disability Index is the most commonly used outcome-measure questionnaire for low back pain in a hospital setting. Each section is scored on a 0-5 scale, 5 representing the greatest disability. The index is calculated by dividing the summed score by the total possible score, which is then multiplied by 100 and expressed as a percentage. Thus, for every question not answered, the denominator is reduced by 5. A score of 0-20 reflects minimal disability, 21-40 moderate disability, 41-60 severe disability, 61-80 crippled, and 81-100 bed-bound.

SECONDARY OUTCOMES:
Lumbal Region Joint Range of Motion | 3 week
  we will use Inclinometer.
Modified Schober Test, | 3 week
  Schober's test is a physical examination used in family medicine, physical medicine and rehabilitation, rheumatology to measure the ability of a patient to flex the lower back.
trunk muscle strength (Lafayette manual muscle strength measuring device) | 3 week
  The Lafayette Manual Muscle Tester (MMT) is an ergonomic hand-held device for objectively quantifying muscle strength. Tests are performed with the clinician applying force to the limb of a patient. The objective is for the clinician to overcome or "break" the patient's resistance.
lower body muscle strength (CSMI-Cybex Humac-Norm isokinetic dynamometer) | 3 week
  A CYBEX Isokinetic Test is used to measure the maximum strength of a joint throughout its available range-of-motion (ROM).
trunk muscle endurance | 3 week
  Trunk muscle endurance of the subjects was evaluated using flexor endurance and Sorensen tests.
Balance assessment (BBS, Biodex Medical Systems), | 3 week
  Using this unique device, clinicians can assess neuromuscular control by quantifying the ability to maintain dynamic bilateral and unilateral postural stability on a static or unstable surface. Use any of four test protocols including fall risk, athletic single leg stability, limits of stability and postural stability.
Visual Analogue Scale (VAS) | 3 week
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain.
The Beck Depression Inventory (BDI) | 3 week
  The Beck Depression Inventory (BDI) is a 21-item self-reporting questionnaire for evaluating the severity of depression in normal and psychiatric populations. The Beck Depression Inventory (BDI) is a 21-item, multiple-choice inventory. Respondents are asked to rate each item based on four response choices according to the severity of the symptoms, ranging from the absence of a symptom to an intense level, during the past week. Individual scale items are scored on a 4-point continuum (0=least, 3=most), with a total summed score range of 0-63. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe.
The Pittsburgh Sleep Quality Index (PSQI) | 3 week
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval. Each of the sleep components yields a score ranging from 0 to 3, with 3 indicating the greatest dysfunction. The sleep component scores are summed to yield a total score ranging from 0 to 21 with the higher total score (referred to as global score) indicating worse sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: gamze demircioğlu, phd(c), Principal Investigator — istanbul medipol hastanesi
Locations (1):
- Gamze Demircioglu, Istanbul, Istanbul Avrupa Kitasi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: data — http://pubmed.ncbi.nlm.nih.gov/30311715/ — Chakravarthy KV, Xing F, Bruno K, Kent AR, Raza A, Hurlemann R, Kinfe TM. A Review of Spinal and Peripheral Neuromodulation and Neuroinflammation: Lessons Learned Thus Far and Future Prospects of Biotype Development. Neuromodulation. 2019 Apr;22(3):235-243. doi: 10.1111/ner.12859. Epub 2018 Oct 12. PMID: 30311715.